CLINICAL TRIAL: NCT06179719
Title: Simultaneous EEG-fMRI Study in Healthy Humans During Induction of Propofol Anesthesia to Investigate the Dynamics of Thalamocortical Functional Connectivity in the Alpha Frequency
Brief Title: EEG-fMRI Experiments During Anesthesia Induction With Propofol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PropofolStudyTUM2023
Record Dates: First submitted 2023-11-23; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy controls (Experimental)
  Interventions: Drug: Propofol; Behavioral: visual flickering stimulation at the alpha frequency

INTERVENTIONS:
Drug: Propofol — Anesthesia will be induced intravenously using the hypnotic drug propofol. The drug is used regularly in everyday clinical practice to carry out general anesthesia, and the intended concentrations are within the usual clinical dosage range. Propofol will be applied via target-controlled infusion (TCI) with a perfusor using TCI set to effect mode as described by Schnider (Schnider et al., 2016). Starting at low concentrations, the effect site concentration will be increased stepwise to achieve the target level of sedation as measured by the Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scale. We aim for three different levels of sedation: low (MOAA/S=5-4), mid (MOAA/S=3-2) and high (MOAA/S=1).
Behavioral: visual flickering stimulation at the alpha frequency — Participants will receive visual stimulation as a flickering light during the different sedation levels, including wakefulness pre- and post-anesthesia. Stimulation will be done with eyes closed in all conditions.

SUMMARY:
This observational study aims to investigate healthy cortical and subcortical neural processes involved in generating intrinsic alpha oscillations during induction of general anesthesia with propofol. To do this, the investigators have designed a simultaneous electroencephalogram (EEG)- MRI (functional MRI and Spectroscopy) experiment with a visual stimulation paradigm that addresses the subject's specific intrinsic alpha rhythm during anesthesia and wakefulness. The main question it aims to answer is: could the investigators address the alpha oscillation system of the healthy brain with external stimulation during anesthesia? This experiment could lead to a better understanding of the mechanisms underlying the generation of alpha oscillations. It could open new doors to diagnostic and treatment options for diseases where alpha oscillations, such as post-operative delirium, seem to be affected.

DETAILED DESCRIPTION:
This study aims to investigate healthy cortical and subcortical neural processes during induction of general anesthesia with propofol, which is clinically relevant for postoperative delirium, a common cognitive disorder, after surgical intervention in the elderly.

Intrinsic neural oscillations within the alpha frequency band (~8-13Hz) can be measured with the EEG, showing the highest power (i.e., amplitude) in occipital electrodes during eyes-closed wakefulness resting state. Under general anesthesia, especially with propofol, the power of these oscillations decreases in the occipital cortex but increases in the frontal cortex. Although neither the exact mechanisms underlying the generation of alpha oscillations nor their dynamics under anesthesia are entirely understood, it has been suggested that the thalamus might be a key player modulating the shift of alpha-band power throughout the brain.

Post-operative delirium (POD) is a complication after a surgical intervention characterized by an acute impairment of consciousness, attention, and arousal with a fluctuating evolution. This is prevalent mainly in elderly patients, especially in those with pre-existing neurocognitive disorders, neurodegenerative disease, and those undergoing complex or emergency procedures. Despite the functional and economic burden this disorder places on the patient and the health system, e.g., it increases hospital stay and risk of mortality, treatment options and risk management strategies are still limited. Several of our previous studies and those from other groups have highlighted the link between alpha oscillations and clinical outcomes related to POD. For instance, low frontal alpha power - both during maintenance and emergence from general anesthesia - is associated with a higher risk of POD. Low frontal alpha power is also associated with pre-operative neurocognitive impairment, a well-described risk factor for POD. The biochemical nature of this association is still unknown; the role of the cholinergic system as a mediator has been suggested.

Therefore, a better understanding of the mechanisms underlying the generation of alpha oscillations and their dynamics under general anesthesia could open new doors to diagnostic and treatment options for POD.

Based on our past EEG-fMRI experiments in healthy subjects applying visual stimulation at the alpha frequency, the investigators have shown that (i) visual stimulation using a rhythmic flickering light at a specific frequency evokes a reliable response in the occipital brain, which can be measured with EEG and functional resonance magnetic imaging (fMRI), (ii) the response to this stimulation can be evaluated via evoked potential/power/coherence analyses (EEG) or functional connectivity analyses (fMRI), and (iii) visual flicker stimulation at/near to a subject's intrinsic alpha frequency, known as the 'individual alpha frequency' (IAF), generates a response within brain areas beyond the occipital cortex, such as frontal and parietal regions and most importantly, the thalamus, suggesting an interaction with - and a method to assess - intrinsic alpha oscillations.

The investigators propose a simultaneous EEG-fMRI study in which young, healthy participants, anesthetized with propofol, are presented with a visual flicker stimulation paradigm at/around the participant's IAF. Our experimental design includes recordings before the participant is anesthetized (wakefulness pre-anesthesia) and during three different anesthesia concentrations (low, mid, and deep). Functional magnetic resonance spectroscopy will be acquired during resting state throughout all states. A wakefulness post-anesthesia recording in resting state without stimulation is also planned. This approach has several advantages. For instance, the simultaneous acquisition makes it possible to correlate the dynamics of alpha oscillations measured by EEG while having access to a whole-brain resolution via fMRI, including subcortical areas like the thalamus. This is relevant to understanding the interaction between cortical and subcortical neural processes generating alpha oscillations.

Furthermore, it exploits the fact that our modality of stimulation at the IAF enhances intrinsic alpha processes, which can potentially become a treatment to reduce the risk of POD under anesthesia. Furthermore, by acquiring functional spectroscopy data, the investigators can detect biochemical changes in the brain during each state. Finally, our experimental design enables, first, a chronologic follow-up of alpha dynamics during the induction of propofol anesthesia, and second, by acquiring data after the intervention, investigators will have an immediate control to contrast before and after anesthesia.

For our participant's safety, propofol anesthesia will be titrated until deep concentrations without eliciting a burst suppression state, avoiding intubation and artificial respiration support.

This study represents an essential step towards understanding alpha oscillatory processes in the awake and anesthetized brain relevant to the future development of potential preventative/treatment options for POD.

ELIGIBILITY:
Inclusion Criteria:

* Female and male healthy individuals (ASA I: assessed according to the American Society of Anesthesiologists Physical Status Classification System a non-acute or chronic disease), non-pregnant, non-smokers, non-drug-users, and presenting no or minimal alcohol use.
* Age: 18 to 35 years
* Capacity to give consent
* Written consent after detailed information.

Exclusion criteria:

* Individuals who do not meet all inclusion criteria
* Previous brain surgery
* History of epileptic seizures
* History of psychiatric or neurological disease
* Physical status other than American Society of Anesthesiologists physical status I, e.g., presence of severe internal or systemic disease
* Chronic intake of medication or drugs (Alcohol, Marihuana, Cocaine, Opioids, Benzodiazepine, etc.)
* Impaired hearing or presence of deafness
* Absence of fluency in the German language
* Known disposition to malignant hyperthermia
* Previous diagnosis of hepatic porphyria
* Body mass index greater than 30 kg/m2
* Gastrointestinal disorders with a disposition for gastroesophageal regurgitation
* Known or suspected difficult airway
* Known hypersensitivity to propofol or any propofol injectable emulsion components (i.e., eggs, eggs products, soybeans, or soy products)
* Atopy/severe allergies/asthma
* Cardiological abnormalities: torsades de pointes, prolonged QT interval, QT changes present since birth.
* Contraindications to MRI (e.g., pacemakers, artificial heart valves, cardioseal, aneurysm clips, implanted magnetic metal parts (screws, plates from surgery), cochlear implants, metal splitters/grenade splinters, acupuncture needle, insulin pump, piercings that cannot be removed, etc)
* Pregnancy
* Subjects with claustrophobia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Visual stimulation at the intrinsic alpha frequency will be related to a change in synchronization in the EEG compared to flankers across all conditions (i.e., wakefulness pre-anesthesia and propofol sedation at low, mid, and high concentrations. | 12 months
  Before propofol sedation administration during resting eyes closed baseline recordings and during the different propofol sedation levels, the investigators expect to see changes in EEG-based oscillatory responses to visual flicker stimulation at the baseline intrinsic alpha frequency compared to control flanker frequencies. These changes imply an interaction between the intrinsic alpha oscillations and the flicker stimulation.
Visual stimulation at the intrinsic alpha frequency will elicit a change in functional connectivity between the thalamus and the cortex during wakefulness as well as during the different propofol sedation levels as compared to flanker frequencies. | 12 months
  During resting baseline conditions (i.e., before propofol sedation administration), the investigators expect a change of functional connectivity between occipitoparietal areas and the thalamus as well as in connectivity between occipitoparietal areas as well as the thalamus and frontal brain areas. With increasing propofol sedation, the investigators expect this selective change in connectivity to intrinsic alpha frequency flicker versus flanker frequencies to diminish.
The change of thalamocortical connectivity mediates the intrinsic alpha frequency-elicited synchronicity changes across modalities (EEG and fMRI) | 12 months
  Concurrent analysis of EEG and fMRI: During resting baseline conditions (i.e., before propofol sedation administration), the investigators expect the phase coupling based on imaginary coherence of alpha oscillations to covary with functional connectivity from fMRI for intrinsic alpha frequency flicker across stimulation repetitions. The investigators expect the supporting brain regions of covarying connectivity across modalities to be centered in the thalamus. With increasing propofol sedation (going from low, mid until high propofol level measured by MOAAS), the investigators expect this cross-modality covariation of connectivity measures for intrinsic alpha frequency flicker frequencies to change.
Choline concentrations in the occipital cortex will change with propofol sedation | 12 months
  The investigators expect choline concentration in the occipital cortex to change with increasing concentrations of propofol sedation.
Intrinsic alpha frequency-elicited synchronicity across modalities (EEG and fMRI) is associated with changes in choline concentrations | 12 months
  Integration of derived measures: The investigators expect both phase coupling of alpha oscillations from EEG as well as changes in thalamocortical functional connectivity in response to visual flicker stimulation at the intrinsic alpha frequency to correlate with changes in choline concentrations measured by Spectroscopy in the occipital cortex.
Simultaneous changes of the aperiodic component of EEG with the different levels of propofol sedation: aperiodic activity in EEG is a potential marker of arousal | 12 months
  The investigators hypothesize that the slope of the aperiodic 1/f distribution will change with increasing levels of propofol sedation across subjects.

SECONDARY OUTCOMES:
Propofol sedation changes the correlation between the global grey matter fMRI blood oxygen level dependent (BOLD) and CSF flow signals. | 12 months
  About a decade ago, a novel mechanism explaining how the brain clears out waste products was postulated (Iliff et al., 2012). This is known as the 'glymphatic hypothesis', and it consists of the transportation of waste products from the brain parenchyma to the periphery facilitated by a continuous circulation of cerebral spinal fluid (CSF flow) throughout the brain (Habilitz & Nedergaad 2021). One driving mechanism of this continuous flow of CSF is global brain activity. The investigators aim to study the effect of propofol anesthesia on the correlation between the global grey matter BOLD and CSF flow signal derived from resting-state fMRI measurements. This idea comes from recent high-impact publications showing first, that during deep sleep, these two signals are highly coupled (Fultz et al., 2019), and second, that this coupling is reduced during neuropsychiatric diseases such as Alzheimer's disease (Han et al., 2021).

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Klinikum rechts der Isar - Klinik für Anästhesiologie und Intensivmedizin, Munich, Bavaria
  - Technische Universität München, München, München (Stadt)

REFERENCES:
- [Background] Iliff JJ, Wang M, Liao Y, Plogg BA, Peng W, Gundersen GA, Benveniste H, Vates GE, Deane R, Goldman SA, Nagelhus EA, Nedergaard M. A paravascular pathway facilitates CSF flow through the brain parenchyma and the clearance of interstitial solutes, including amyloid beta. Sci Transl Med. 2012 Aug 15;4(147):147ra111. doi: 10.1126/scitranslmed.3003748. PMID 22896675
- [Background] Hablitz LM, Nedergaard M. The Glymphatic System: A Novel Component of Fundamental Neurobiology. J Neurosci. 2021 Sep 15;41(37):7698-7711. doi: 10.1523/JNEUROSCI.0619-21.2021. PMID 34526407
- [Background] Fultz NE, Bonmassar G, Setsompop K, Stickgold RA, Rosen BR, Polimeni JR, Lewis LD. Coupled electrophysiological, hemodynamic, and cerebrospinal fluid oscillations in human sleep. Science. 2019 Nov 1;366(6465):628-631. doi: 10.1126/science.aax5440. PMID 31672896
- [Background] Han F, Chen J, Belkin-Rosen A, Gu Y, Luo L, Buxton OM, Liu X; Alzheimer's Disease Neuroimaging Initiative. Reduced coupling between cerebrospinal fluid flow and global brain activity is linked to Alzheimer disease-related pathology. PLoS Biol. 2021 Jun 1;19(6):e3001233. doi: 10.1371/journal.pbio.3001233. eCollection 2021 Jun. PMID 34061820